CLINICAL TRIAL: NCT03412175
Title: CREATION Health Lifestyle Intervention
Acronym: CHLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 878401
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Risk
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): Participants in the lifestyle intervention arm will receive 6 individual visits with a CREATION Health Specialist over a 3 month period, and one follow up visit at 6 months. The visits include one 2 hour-long initial assessment, four 60-minute motivational interview sessions, and two 60-minute reassessments. Visits will focus on tailoring the intervention care plan to each individual, goal-setting, action plans, self-monitoring, identification of personal and social barriers to change, self-regulatory techniques, and provision of psychosocial support using motivational interviewing techniques.
  Interventions: Behavioral: Behavioral Intervention
- Control Group (No Intervention): Participants in the control group will receive usual care as provided by their primary care physician. Participants in the control group will complete biometrics, surveys, and assessments at Visits 0, 5 and 6.

INTERVENTIONS:
Behavioral: Behavioral Intervention — The CREATION Health Specialist (CHS) will review with the participant his/her biometrics, assessments, and surveys. The CHS will identify the participant's strengths and weaknesses thereby tailoring the intervention care plan to the participant. Together the participant and CHS will work on goal-setting, action plans, self-monitoring, identification of personal and social barriers to change, and self-regulatory techniques.
  Arms: Behavioral Intervention

SUMMARY:
The CREATION Health Lifestyle Intervention (CHLI) will study the effect of a lifestyle intervention program on the cardiovascular risk profile (blood pressure, BMI, and Hemoglobin A1C) of participants diagnosed with hypertension and/or type 2 diabetes.

DETAILED DESCRIPTION:
The CREATION Health Lifestyle intervention is targeted at improving the cardiovascular risk profiles (blood pressure, BMI, and Hemoglobin A1C) of participants diagnosed with hypertension and/or type 2 diabetes. The intervention is designed to address the whole person and is based on the CREATION Health framework. Participants in the lifestyle intervention arm will receive 6 individual visits with a CREATION Health Specialist over a 3 month period, and one follow up visit at 6 months. The visits include one 2 hour-long initial assessment, four 60-minute motivational interview sessions, and two 60-minute reassessments. Visits will focus on tailoring the intervention care plan to each individual, goal-setting, action plans, self-monitoring, identification of personal and social barriers to change, self-regulatory techniques, and provision of psychosocial support using motivational interviewing techniques. Using the CREATION Health framework, the CREATION Health Specialist will educate the participant and make recommendations for lifestyle modifications that lead to reduction in cardiovascular disease risk by focusing on: reduced energy intake, primarily via lowering fat intake to <30% of caloric intake; increased physical activity to 150 minutes per week; smoking cessation; limited sodium intake; and limited alcohol intake.

Intervention fidelity will be determined by tracking the content of visits on encounter forms. There will also be a quality assurance assessment by audio-taping a select number of CHS-patient visits. The audiotapes will be reviewed by the study team and CHS for adherence to study intervention protocols.

Participants in the intervention group will also receive a health journal to document progress and a CREATION Health workbook that introduces the CREATION Health framework in more detail. The workbook explains each concept of the CREATION Health framework: Choice; Rest; Environment; Activity; Trust in God; Interpersonal relationships; Outlook; and Nutrition. Participants in the intervention group will receive a CREATION Health One-sentence Journal.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 2 Diabetes, fasting glucose >125, or Hg A1C >6.5% and/or
2. Diagnosis of Hypertension
3. Age 18 or older
4. Agree to participate in all aspects of study intervention and assessments
5. Able to give informed consent
6. Access to home phone or mobile phone

Exclusion Criteria:

1. Current use of oral corticosteroids
2. Current use of psychotropics for psychosis or bipolar disorder
3. Use of weight-loss medication in the past 3 months
4. Psychiatric hospitalization in the past 3 years
5. Cancer diagnosis or treatment in the past 3 years
6. History of MI, CABG, stroke, PTCA, balloon pump, etc in past 2 years
7. Hemoglobin A1C 12% or more on two occasion in the past 6 months
8. Pregnancy
9. Severe debilitating medical condition that would interfere with completion of intervention
10. Unable to speak, read, and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 6 months
  A 6 mm Hg reduction in systolic blood pressure/diastolic blood pressure as measured in clinic in participants diagnosed with Hypertension
Hemoglobin A1C | 6 months
  A reduction of Hemoglobin A1C in participants diagnosed with Type II Diabetes Mellitus to less than 6% as measured by fasting blood work

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Robinson, Principal Investigator — Center for CREATION Health Research
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Executive Summary: Heart Disease and Stroke Statistics--2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):447-54. doi: 10.1161/CIR.0000000000000366. No abstract available. PMID 26811276
- [Background] Spring B, Ockene JK, Gidding SS, Mozaffarian D, Moore S, Rosal MC, Brown MD, Vafiadis DK, Cohen DL, Burke LE, Lloyd-Jones D; American Heart Association Behavior Change Committee of the Council on Epidemiology and Prevention, Council on Lifestyle and Cardiometabolic Health, Council for High Blood Pressure Research, and Council on Cardiovascular and Stroke Nursing. Better population health through behavior change in adults: a call to action. Circulation. 2013 Nov 5;128(19):2169-76. doi: 10.1161/01.cir.0000435173.25936.e1. Epub 2013 Oct 7. No abstract available. PMID 24100544
- See also: Centers for Medicare and Medicaid Services. Decision Memo for Intensive Behavioral Therapy for Obesity. Website. [cited 2016 February 4]. — https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?&NcaName=Intensive%20Behavioral%20Therapy%20for%20Obesity&bc=ACAAAAAAIAAA&NCAId=253&